CLINICAL TRIAL: NCT06024772
Title: Prostate Cancer Diagnosis by Multiparametric Ultrasound (Clinical)
Brief Title: Multiparametric Ultrasound for the Diagnosis of Clinically Significant Prostate Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Eindhoven University of Technology (Other); Eigen (Other); GE Healthcare (Industry)
Responsible Party: Principal Investigator, Flemming Forsberg, Professor - Radiology, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: iRISID-2022-1191; JT 20767 (Other: JeffTrial Number)
Record Dates: First submitted 2023-08-18; First posted 2023-09-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — perflutren; Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (mp-MRI, Definity, mp-US, prostate biopsies) (Experimental): Patients undergo mp-MRI, receive Definity IV, and undergo transrectal mp-US and prostate biopsies on study.
  Interventions: Procedure: ultiparametric Magnetic Resonance Imaging; Drug: Perflutren lipid microsphere; Procedure: Transrectal Ultrasound; Procedure: Biopsy of Prostate

INTERVENTIONS:
Procedure: ultiparametric Magnetic Resonance Imaging — Undergo mp-MRI
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI
Drug: Perflutren lipid microsphere — Given IV
  Other Names: Definity
Procedure: Transrectal Ultrasound — Undergo transrectal mp-US
  Other Names: endorectal ultrasound; ERUS; TRUS
Procedure: Biopsy of Prostate — Undergo prostate biopsies
  Other Names: Prostate Biopsy; Prostatic Biopsy

SUMMARY:
This phase III trial compares the use of contrast-enhanced multiparametric ultrasound (mp-US) to multiparametric magnetic resonance imaging (mp-MRI) for the diagnosis of clinically significant prostate cancer (PCa). A mp-US is a procedure in which a probe that sends out high-energy sound waves is inserted into the rectum. The sound waves are bounced off internal tissues or organs and make echoes. The echoes form a picture of body tissue called a sonogram. Perflutren lipid michrosphere (Definity) is a contrast agent that uses microbubbles to enhance ultrasound images of the prostate. Doctors hope to learn if the Definity-enhanced mp-US imaging technique can accurately direct targeted biopsy for the detection of clinically significant prostate cancer when compared to standard of care mp-MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate non-inferiority between the detection rate of clinically significant PCa with 3-dimensional (3D) mp-US + systematic biopsy compared to the detection rate of mp-MRI + systematic biopsy.

II. To compare the positive yield of targeted biopsy cores based on mp-US + systematic biopsy with targeted biopsy based on mp-MRI + systematic biopsy, for detection of clinically significant PCa.

SECONDARY OBJECTIVES:

I. To demonstrate non-inferiority of a biopsy approach utilizing targeted biopsy cores based on mp-US compared with targeted biopsy based on mp-MRI, for detection of clinically significant PCa.

II. To construct an optimal logistic regression model to predict the presence of clinically significant PCa based on the mp-US elements as well as the prostate specific antigen (PSA), PSA velocity and any other biological variables (e.g., age).

OUTLINE:

Patients undergo mp-MRI, receive Definity intravenously (IV), and undergo transrectal mp-US and prostate biopsies on study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be scheduled for a prostate biopsy, based on an elevated PSA (> 3.0ng/ml) per most recent National Comprehensive Cancer Network (NCCN) guidelines, elevated PSA velocity (> 0.75ng/ml/year), or abnormal digital rectal examination
* Subject must be able and willing to give written informed consent for a contrast enhanced ultrasound study of the prostate including the additional study biopsies
* Subject must be a male at least 18 years of age when informed consent is obtained

Exclusion Criteria:

* Participant in a clinical trial involving an investigational drug within the past 30 days
* Patients with known or suspected hypersensitivity to perflutren, polyethylene glycol (PEG), or any other component of Definity
* Previous treatment for prostate cancer, including hormone therapy
* Clinically unstable, severely ill, or moribund as per treating physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer (PCa) detection rate of 3-dimensional (3D) multiparametric ultrasound (mp-US) combined with systematic biopsy | Up to 2 years
  Will compare PCa detection rate of 3D mp-US combined with systematic biopsy to detection rate of multiparametric magnetic resonance imaging (mp-MRI) combined with systematic biopsy. Will evaluate paired biopsy data for non-inferiority and superiority endpoints, comparing the detection rate of clinically significant PCa with mp-US + systematic biopsy to the detection rate of mp-MRI + systematic biopsy. This analysis will be repeated using both definitions of clinically significant PCa. Categorical data will be summarized as counts and percentages (or proportions) and continuous data will be summarized with descriptive statistics such as mean, standard deviation (SD), median, and range.

SECONDARY OUTCOMES:
PCa detection rate of 3D mp-US | Up to 2 years
  Categorical data will be summarized as counts and percentages (or proportions) and continuous data will be summarized with descriptive statistics such as mean, SD, median, and range. Continuous data will be analyzed using t-tests, or log-rank tests if data are not normally distributed. Variance is expressed through 95% confidence intervals and a significance level of 5% with Bonferroni correction for multiple comparisons will be used to control the group-wise error of the study for individual comparisons.
Accuracy of PCa detection by biopsy using the optimal logistical model based around mp-US compared to the optimal logistical model based around mp-MRI | Up to 2 years
  Will evaluate the accuracty of the optimal logistic model combining the mp-US elements as well as the prostate specific antigen, prostate specific antigen velocity and other biological variables.

CONTACTS AND LOCATIONS:
Locations (2):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States
- Amsterdam Medical Center, Amsterdam-Zuidoost, Netherlands